CLINICAL TRIAL: NCT07229781
Title: Glycemic Effects of a Mediterranean-Style Dietary Pattern Containing Potatoes in Adults With Prediabetes
Brief Title: Mediterranean Diet and Blood Sugar Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Alliance for Potato Research & Education (Unknown)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MDP
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Prediabetes
Keywords: prediabetes; diet; nutrition; Mediterranean diet; cardiovascular disease
MeSH Terms: conditions — Prediabetic State; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean-style diet with potato (MED-P) (Experimental): Mediterranean-style diet that includes 1 medium potato/day/2000 kcal replacing some grains
  Interventions: Other: Mediterranean-style diet with potatoes
- Traditional-style Mediterranean dietary pattern (MED) (Active Comparator): A traditional-style Mediterranean diet that does not contain potatoes (potatoes are not a defining feature of this diet) and is higher in grains.
  Interventions: Other: Traditional-style Mediterranean diet

INTERVENTIONS:
Other: Mediterranean-style diet with potatoes — The diet will contain 1 medium potato/day/2000 kcal
  Arms: Mediterranean-style diet with potato (MED-P)
Other: Traditional-style Mediterranean diet — Traditional-style Mediterranean diet higher in grains
  Arms: Traditional-style Mediterranean dietary pattern (MED)

SUMMARY:
The purpose of this research study is to determine if a healthy Mediterranean diet containing one medium potato/day has equivalent or non-different effects on risk factors for type 2 diabetes and heart disease compared to a healthy Mediterranean diet without potatoes in adults with prediabetes. Participants will be randomly assigned to one of the test diets and be asked to consume this diet for 12 weeks (84 days). Testing will be conducted at the beginning and end of the study.

DETAILED DESCRIPTION:
This is a 12-week, 2-arm parallel, randomized controlled feeding trial. Participants will be randomized to either a Mediterranean-style diet that includes 1 medium potato/day/2000 kcal replacing some grains , or a traditional-style Mediterranean dietary pattern without potatoes. All food will be provided for the 12-week study duration.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-65 years
* Prediabetes assessed by an HbA1c of 5.7-6.4% or fasting glucose 100-125 mg/dL at screening
* BMI 25-40 kg/m2 at screening

Exclusion Criteria:

* HbA1c ≥6.5% at screening
* LDL-C (calculated with the Martin-Hopkins equation) ≥190 mg/dL at screening
* Hemoglobin <13.2 g/dL at screening
* Fasting triglycerides >350 mg/dL at screening

  -≥10% change in body weight within the 6 months prior to enrollment
* Blood pressure >140/90 mmHg at screening
* Type 1 or type 2 diabetes
* Prescription of anti-hypertensive, lipid-lowering, or glucose-lowering drugs
* Intake of supplements that affect the outcomes of interest (i.e., lipid, blood pressure, or glucose lowering; vitamin C or multi-vitamins containing vitamin C) and are unwilling to cease during the study period.
* History of liver, kidney, or autoimmune disease
* Prior cardiovascular event (e.g., stroke, heart attack)
* Current pregnancy or intention of pregnancy within the next 6 months
* Lactation within the prior 6 months
* Allergy/intolerance/sensitivity/dislike of any foods in the study menus
* Antibiotic use within the prior 1 month
* Oral steroid use within the prior 1 month
* Use of tobacco or nicotine-containing products within the past 6 months
* History of cancer at any site within the past 10 years (eligible if ≥10 years without recurrence) or non-melanoma skin cancer within the past 5 years (eligible if ≥5 years without recurrence)
* Participation in another clinical trial within 60 days of baseline
* Currently following a restricted or weight-loss diet
* Prior bariatric surgery
* Intake of >14 alcoholic drinks/week and/or not willing to avoid alcohol consumption for 48 hours prior to test visits
* Principal Investigator discretion related to the potential participant's ability to adhere to the study requirements, including being able to come to attend visits
* Does not speak and/or understand English
* Unwilling to refrain from donating blood during the study
* Weight <110 lb

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 12-weeks
  HbA1c will be assessed at baseline and 12-weeks and expressed as percentage . The change in HbA1c will be calculated by subtracting the baseline value from the 12 week value and expressed as percentage point change.

SECONDARY OUTCOMES:
Change in fasting glucose | 12-weeks
  Change in fasting plasma glucose expressed as mg/dL. Change in glucose will be calculated as the mean of the 12 week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in mean glucose | 12-weeks
  Change in mean glucose assessed by a continuous glucose monitor (CGM) expressed as mg/dL. Change in mean glucose will be calculated as mean glucose assessed from 7 days of CGM wear at 12 weeks minus mean glucose assessed from 7 days of CGM wear at baseline.
Change in mean time in range | 12-weeks
  Change in mean time in range (glucose 70-140 mg/dL) assessed by a continuous glucose monitor (CGM) expressed as minutes per day. Change in mean time in range will be calculated as mean time in range assessed from 7 days of CGM wear at 12 weeks minus mean time in range assessed from 7 days of CGM wear at baseline.
Change in glycemic variability | 12-weeks
  Change in mean glycemic variability assessed by a continuous glucose monitor (CGM) expressed as the coefficient of variability. Change in mean glycemic variability will be calculated as mean glycemic variability assessed from 7 days of CGM wear at 12 weeks minus mean glycemic variability assessed from 7 days of CGM wear at baseline.
Change in fasting insulin | 12-weeks
  Change in fasting serum insulin expressed as micro IU/mL. Change in insulin will be calculated as the mean of the 12 week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in homeostatic model of insulin resistance (HOMA-IR) | 12-weeks
  Homeostatic model of insulin resistance (HOMA-IR) will be calculated from insulin and glucose measured from a fasting blood sample. Calculated as (insulin × glucose) / 22.5. Change in HOMA-IR will be calculated as the mean of the 12 week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in LDL-Cholesterol | 12-weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in LDL-cholesterol will be calculated as the mean of the 12-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in apolipoprotein B | 12-weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in apolipoprotein B will be calculated by subtracting the baseline value from the 12 week value.
Change in non-HDL cholesterol | 12-weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in non-HDL cholesterol will be calculated as the mean of the 12-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in Total Cholesterol | 12-weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in total cholesterol will be calculated as the mean of the 12-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in HDL-Cholesterol | 12-weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in HDL-cholesterol will be calculated as the mean of the 12-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in Triglycerides | 12-weeks
  Assessed from fasting blood draw expressed in mg/dL. Change in triglycerides will be calculated as the mean of the 12-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in C-reactive protein | 12-weeks
  Assessed from fasting blood draw expressed in mg/L. Change in C-reactive protein will be calculated as the mean of the 12-week measures (i.e., mean of day 1 and day 2 values) minus the mean of the baseline measures (i.e., mean of day 1 and day 2 values).
Change in Central Systolic and Diastolic Blood Pressure | 12-weeks
  Central blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical) at baseline & 12 weeks. Change will be calculated by subtracting the baseline value from the end point value.
Change in Peripheral Systolic and Diastolic Blood Pressure | 12-weeks
  Peripheral blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical) at baseline & 12 weeks. Change will be calculated by subtracting the baseline value from the end point value.
Change in Carotid-Femoral Pulse Wave Velocity | 12-weeks
  Measured assessed using a SphymoCor Xcel (Atcor Medical) at baseline & 12 weeks. Change will be calculated by subtracting the baseline value from the end point value.
Change in particle size and number of LDL, HDL, triglyceride rich lipoproteins | 12-weeks
  Measured via Nuclear Magnetic Resonance
Diet Satisfaction | 12-weeks
  Participants will complete a survey that we have previously developed to assess diet satisfaction at 12 weeks.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: The SAP and protocol will be posted on clinicaltrials.gov prior to enrollment commencing.